CLINICAL TRIAL: NCT07152743
Title: L'Esperienza Del Padre e Della Madre in Relazione Alla Presenza Del Padre All'Evento Parto in Caso di Taglio Cesareo Programmato: Uno Studio Qualitativo Fenomenologico
Brief Title: The Experience of Fathers and Mothers in Relation to the Presence of the Father at the Birth in the Case of a Planned Caesarean Section: a Qualitative Phenomenological Study
Acronym: "PARENTS"
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Preziosi Jessica, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7528
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Cesarean Section; Parturition
Keywords: Parent; Father; Cesarean Section

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pregnancy and childbirth represent a crucial transition for couples, involving significant psychological and emotional adaptation. The World Health Organization recommends that all women have the possibility to be accompanied by a support person of their choice during labor and birth. The presence of a trusted companion can provide emotional reassurance, improve communication with health professionals, and support non-pharmacological pain management, often reducing the need for medical interventions.

Fathers who attend childbirth frequently describe their participation as a meaningful and positive experience, strengthening their relationship with both the mother and the newborn. However, in the case of elective cesarean section, the father's presence in the operating room is not always allowed, especially when there is a high risk of complications (such as major hemorrhage). This variability may influence how mothers and fathers experience the birth.

This qualitative, single-center, non-funded study aims to explore and describe the lived experiences of mothers and fathers regarding the presence or absence of the father during an elective cesarean section.

After informed consent, couples will be invited to participate in a semi-structured interview conducted 48-72 hours after birth, during postpartum hospitalization at Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome. The interview, lasting approximately 20-30 minutes, will be audio-recorded and anonymized. Participants may withdraw at any time without consequences for their care.

The primary objective is to describe the experience of both mothers and fathers in relation to whether the father was present or absent at the birth. Secondary objectives include:

describing demographic and obstetric characteristics of participating women,

exploring expectations and emotions of fathers who attended the cesarean birth and of their partners,

exploring the experiences of fathers who could not be present, and of their partners,

evaluating the perceived support provided by healthcare staff,

identifying unexpected needs or desires expressed by participants.

A purposive sample of approximately 30 couples will be recruited (15 where the father is present and 15 where he is absent). Recruitment will continue until data saturation is reached. Data will be analyzed using thematic analysis, following established qualitative research methods.

This study will provide new insights into how the presence or absence of the father during elective cesarean section shapes the birth experience for both parents. The results may support policies and practices aimed at improving emotional well-being, strengthening family bonds, and enhancing the quality of maternity care.

ELIGIBILITY:
Inclusion Criteria:

* Women who have undergone an elective cesarean section
* Women who have provided written informed consent
* Women with gestational age > 37 weeks + 0 days

Exclusion Criteria:

* Fathers or mothers under 18 years of age
* Fathers or mothers unable to read and understand the Italian language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Couples (mother and father) experiencing an elective cesarean section at Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy. Mothers must be ≥37 weeks gestation and have provided written informed consent. Fathers and mothers must be ≥18 years old and able to understand Italian.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To describe the lived experience of mothers and fathers in relation to the father's presence or absence during elective cesarean birth. | 48-72 hours postpartum
  Semi-structured interview conducted with mothers and fathers after childbirth